CLINICAL TRIAL: NCT06497283
Title: The Effect of Intraoperative Binaural Sound on Remifentanil Dose Required for General Anesthesia Using Remimazolam: a Randomized, Placebo-controlled Trial
Brief Title: Binaural Sound for Remimazolam Maintenance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Chang Kim, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 3-2024-0171
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: General Anesthesia; Prostate Cancer Stage; Uterine Myoma
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I (Binaural) (Experimental): Binaural sound using earphone will be applied.
  Interventions: Procedure: Binaural sound
- II (Placebo) (Placebo Comparator): Only headphone without sound will be applied.
  Interventions: Procedure: Binaural sound

INTERVENTIONS:
Procedure: Binaural sound — Binaural sound: Binaural sound will be applied.

SUMMARY:
It is important to decrease the remifentanil dose for general anesthesia maintenance when using remimazolam. We will evaluate the effect of binaural sound on general anesthesia maintenance with remimazolam infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for general anesthesia
2. Patients aged 20-60
3. Patients with American Society of Anesthesiologist physical status classification 1-2
4. Patients with ideal body weight 50-80 kg

Exclusion Criteria:

1. Patients with hearing disability
2. Patients using opioids or sedatives in 1 week
3. Patients who are dependent for alcoholics or drugs
4. Patients with hypersensitivities to remimazolam or remifentanil
5. Patients with arrhythmia, cardiovascular disease, heart failure, or hypovolemia
6. Patients with liver failure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Intraoperative remifentanil dose | At anesthesia day 0
  Intraoperative remifentanil dose will be measured at anesthesia day 0.

SECONDARY OUTCOMES:
Intraoperative remimazolam dose | At anesthesia day 0
  Intraoperative remimazolam dose will be measured at anesthesia day 0.
Pain score (0:no pain, 10:maximal pain) | At anesthesia day 0 and 1
  Pain score (0:no pain, 10:maximal pain) will be measured at anesthesia day 0 and 1.
Electroencephalography | At anesthesia day 0
  The relative power of alpha, beta, delta, gamma, and theta band in electroencephalography will be measured at anesthesia day 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea